CLINICAL TRIAL: NCT01742598
Title: Assessment of St Jude Medical Portico Re-sheathable Transapical Aortic Valve System
Acronym: Portico TA EU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1106
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Severe Symptomatic Aortic Stenosis
Keywords: TAVI; TAVR; aortic stenosis; Transcatheter; valvular heart disease; aortic valve stenosis; aortic valve replacement; transcatheter aortic valve implantation
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Portico Implant (Experimental)
  Interventions: Device: Portico Transapical Aortic Valve System

INTERVENTIONS:
Device: Portico Transapical Aortic Valve System

SUMMARY:
The purpose of this study is to assess the safety and performance of the 23mm Portico Transcatheter Heart Valve and the TAVI Transapical Delivery System in subjects with severe symptomatic aortic stenosis

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed the study Informed Consent Form and Data Protection Form prior to participating in the study.
2. Subject is 65 years of age or older at the time of index procedure, and/or has comorbidities that, in the opinion of the Principal Investigator or the Subject Selection Committee, preclude surgical valve replacement.
3. Subject's aortic annulus is 19-21mm diameter as measured by echocardiography (echo) or CT conducted within 90 days prior to the index procedure.
4. Subject has senile degenerative aortic stenosis with echocardiography derived mean gradient greater than (>) 40mmHg or jet velocity greater than 4.0 m/s or an initial valve area of less than (<) 0.8 cm2 (or aortic valve area index less than or equal to (≤) 0.6 cm2/m2). (Baseline measurement taken by echo within 90 days of index procedure).
5. Subject has symptomatic aortic stenosis as demonstrated by NYHA Functional Classification of II, III, or IV.
6. Subject is deemed high operable risk and suitable for TAVI per the medical opinion of the Subject Selection Committee.
7. Subject's predicted operative mortality or serious, irreversible morbidity risk is less than (<) 50% at 30 days post index procedure.

Exclusion Criteria:

1. Subject is unwilling or unable to comply with all study-required follow-up evaluations.
2. Subject has a documented history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within 6 months (less than or equal to (≤) 180 days) prior to the index procedure.
3. Subject has a chest condition than prevents transapical access.
4. Subject has carotid artery disease requiring intervention.
5. Subject has documented evidence of a myocardial infarction (MI) within 6 months (less than or equal to (≤) 180 days) prior to the index procedure.
6. Subject has a native aortic valve that is congenitally unicuspid, bicuspid, quadricuspid or non-calcified as seen by echocardiography.
7. Subject has mitral valvular regurgitation greater than (>) grade III.
8. Subject has moderate or severe mitral stenosis.
9. Subject has aortic root angulation greater than (>) 70 degrees (horizontal aorta).
10. The distance from the left ventricular apex to the aortic annulus is less than (<) 45mm (4.5cm).
11. Subject has a pre-existing prosthetic cardiac device, valve, or prosthetic ring in any position.
12. Subject refuses any blood product transfusion.
13. Subject refuses surgical valve replacement.
14. Subject has left ventricular ejection fraction (LVEF) less than (<) 20%.
15. Subject has documented, untreated symptomatic coronary artery disease (CAD) requiring revascularization.
16. Subject has had a percutaneous interventional or other invasive cardiovascular or peripheral vascular procedure less than or equal to (≤) 14 days of index procedure.
17. Subject has severe basal septal hypertrophy that would interfere with transcatheter valve placement.
18. Subject has a history of, or is currently diagnosed with endocarditis.
19. Subject has imaging evidence of intracardiac mass, thrombus, or vegetation.
20. Subject is considered hemodynamically unstable (requiring inotropic support or mechanical heart assistance).
21. Subject is in acute pulmonary edema or requiring intravenous diuretic therapy to stabilize heart failure.
22. Subject with significant pulmonary disease as determined and documented by the Investigator.
23. Subject has significant chronic steroid use as determined and documented by the Investigator.
24. Subject has a documented hypersensitivity or contraindication to anticoagulant or antiplatelet medication.
25. Subject has renal insufficiency as evidenced by a serum creatinine greater than (>) 3.0 mg/dL (265.5µmol/L) or end-stage renal disease requiring chronic dialysis.
26. Subject has morbid obesity defined as a BMI greater than or equal to (≥) 40.
27. Subject has ongoing infection or sepsis.
28. Subject has blood dyscrasias (e.g., leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy).
29. Subject has a current autoimmune disease that, in the opinion of the Principal Investigator or the Subject Selection Committee, precludes the subject from study participation.
30. Significant ascending aortic disease documented by diameter greater than 40mm.
31. Subject has an active peptic ulcer or has had gastrointestinal (GI) bleeding within 90 days prior to the index procedure.
32. Subject is currently participating in another investigational drug or device study.
33. Subject requires emergency surgery for any reason.
34. Subject has a life expectancy less than (<) 12 months.
35. Subject has other medical, social or psychological conditions that, in the opinion of the Principal Investigator or the Subject Selection Committee, preclude the subject from study participation.
36. Subject is diagnosed with dementia or admitted to a chronic care facility which would fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits.
37. Subject has a documented allergy to contrast media, nitinol alloys, porcine tissue, or bovine tissue.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 30 days

SECONDARY OUTCOMES:
Event rates | 30 days
  * Cardiovascular mortality
  * Myocardial Infarction (MI)
  * Major Stroke
  * Minor Stroke
  * Acute Kidney Injury (AKI)
  * Vascular access site and Access-related complications
  * Bleeding
  * Composite of periprocedural encephalopathy, all stroke, and all TIA
Functional improvements from baseline | 30 days
  * NYHA Functional Classification
  * Six Minute Walk Test
  * Effective Orifice Area (EOA)
Acute device success | At time of procedure
  * Successful apical access, delivery and deployment of the device and successful retrieval of the delivery system,
  * Correct position of the device in the proper anatomical location,
  * Intended performance of the prosthetic heart valve (Aortic Valve Area greater than (>)1.0 cm2 and mean aortic valve gradient less than (<) 20 mmHg or peak velocity less than (<) 3 m/s, without moderate or severe prosthetic valve AR), and
  * Only one valve implanted in the proper anatomical location

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walther, MD, PhD, Principal Investigator — Kerckhoff Klinik
Locations (1):
- King's College Hospital, London, United Kingdom